CLINICAL TRIAL: NCT05937594
Title: Understanding the microRNA Response to Opioid Withdrawal and Their Uses as Potential Biomarkers for Neonatal Abstinence Syndrome
Brief Title: MicroRNA Biomarkers for Neonatal Opioid Withdrawal Syndrome
Status: Recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven Hicks, Associate Professor of Pediatrics, Penn State University
Other Study IDs: 13565; F30DA057094 (NIH)
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Opioid Withdrawal Syndrome; Neonatal Abstinence Syndrome
Keywords: microRNA; saliva; neurodevelopmental; exosomes; infant
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva swab samples are collected from infants. Saliva samples are immediately stored at -80 for later nucleic acid extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants exposed to in utero opiates: Infants that meet IRB-approved inclusion/exclusion criteria.
  Interventions: Genetic: Buccal swab saliva for further genetic testing

INTERVENTIONS:
Genetic: Buccal swab saliva for further genetic testing — Genetic testing. Whole saliva RNA will be isolated for downstream microRNA quantification.

SUMMARY:
Infants with neonatal abstinence syndrome (NAS) experience prolonged hospital stays and poor neurodevelopmental outcomes, in-part because of the lack of accurate, individualized, biologic assessments available to manage this increasingly common medical condition. The proposed study will define the molecular mechanisms that regulate the response to opioid withdrawal in the developing brain by focusing on three candidate microRNAs (let-7a, miR-146a, miR-192) that have been shown to respond to opioid exposure in animal models and adults, and are impacted in both my preliminary study of infants with NAS, and my human neural progenitor cell (NPC) design of opioid withdrawal. By determining the mechanism through which microRNAs impact NPC differentiation in opioid withdrawal, and determining whether exosomal salivary microRNA levels predict treatment dose and neurodevelopmental outcomes in infants with NAS, this study will enhance our knowledge of NAS-related biology and identify potential biomarkers that could improve medical care for this important medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Newborns ≥35weeks gestation with chronic in-utero opioid exposure (>1month of gestation exposure). Maternal exposure will be determined by evaluating the medical records for maternal medication use, maternal urine toxicology and neonatal meconium toxicology results per standard clinical care
* Neonates born at Penn State Hershey Medical Center or transferred at <48 hours after birth
* Mothers with chronic in-utero opioid use during pregnancy ( ≥1month of gestation)

Exclusion Criteria:

* <35 week gestation
* Infant required mechanical ventilation or non-invasive mechanical support
* Infant exposure to magnesium sulfate
* Opioid-exposed neonates who are actively receiving dextrose infusion for persistent neonatal hypoglycemia at the time of enrollment (<48hours after birth).
* Infant with major congenital anomalies
* Parent or guardian unable to provide consent
* Mothers and neonates without history of opioid exposure/dependence

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants enrolled into the study were exposed to opiates in-utero for at least one month of gestation. All infants enrolled meet the eligibility criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcome scores | 6 months of age
  Measured by Ages and Stages Questionnaire-3, score scale 0-60
Maximum concentration of morphine required for withdrawal symptom control | Measured during the course of hospital stay
  Measured in mg/kg/ml
Salivary microRNA level let-7a | Buccal swab collected within 96 hrs of life and at discharge
  Relative fluorescence (Cq) measured by qPCR using established housekeeping gene
Salivary level of microRNA-146a | Buccal swab collected within 96 hrs of life and at discharge
  Relative fluorescence (Cq) measured by qPCR using established housekeeping gene
Salivary level of microRNA-192 | Buccal swab collected within 96 hrs of life and at discharge
  Relative fluorescence (Cq) measured by qPCR using established housekeeping gene
Salivary level of microRNA-149-3p | Buccal swab collected within 96 hrs of life and at discharge
  Relative fluorescence (Cq) measured by qPCR using established housekeeping gene

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Hicks, MD, PhD, Principal Investigator — Associate Professor of Pediatrics
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No